CLINICAL TRIAL: NCT05740514
Title: Targeting Vascular and Skeletal Muscle Health to Improve Quality of Life in Males and Females with Type 1 Diabetes
Brief Title: Healthy Outcomes for Muscle with Exercise in T1D
Acronym: HOME T1D
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Thomas Hawke, Professor, McMaster University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 15516
Record Dates: First submitted 2023-01-25; First posted 2023-02-23 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Study subjects will participate in a twelve-week exercise program. Following this time, a one-week detraining period will ensue. Following this detraining period, study subjects will re-engage in a four-week exercise program.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Twelve-week Exercise (Experimental): Study participants will participate in an exercise program consisting of aerobic and resistance exercise. This arm will last twelve weeks.
  Interventions: Behavioral: Exercise
- One-week Detraining (Experimental): Study participants will undergo unilateral knee immobilization for a one-week period.
  Interventions: Behavioral: De-training
- Four-week Re-training (Experimental): Study participants will once again participate in an exercise program consisting of aerobic and resistance exercise. This arm will last four weeks.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Exercise training.
  Arms: Four-week Re-training; Twelve-week Exercise
Behavioral: De-training — Exercise de-training via unilateral knee immobilization.
  Arms: One-week Detraining

SUMMARY:
Over 300,000 people in Canada suffer from Type 1 Diabetes (T1D), a chronic condition whose incidence rate has been increasing in Canada every year by 5.1% (higher than the global average). While exogenous insulin injections allow those with T1D to live, it is not a cure, and those with T1D develop severe complications (kidney failure, cardiovascular disease). Strategies to regress the development of these complications, minimize healthcare system burden, and save the lives of Canadians are urgently needed.

Undertaking regular exercise is an obvious strategy for those with T1D and has many well-established health benefits. Despite these benefits, adults with T1D exercise less frequently due to fear of severe hypoglycemia and a lack of knowledge of effective exercise strategies. Adding to this complexity, the investigators have recently shown that males and females elicit differential impairments in skeletal muscle metabolism in response to T1D. These differences may extend to the peripheral microvasculature and may lead to sexual dimorphism in the health benefits of exercise for those with T1D. Ultimately, developing a healthy muscle mass, including microvasculature, will help mitigate dysglycemic and dyslipidemic fluctuations and improve insulin sensitivity.

The overarching purpose of this proposed study is to determine the impact of T1D on human skeletal muscle and its microvasculature over the lifespan in males and females, and its responses to exercise training and detraining.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18-30 or 45-65
* Sedentary or recreationally active, as defined by self-reported activity levels below the recommended 150-minute minimum of moderate-to-vigorous intensity physical activity per week

Exclusion Criteria:

* Chronic use of anti-inflammatory, glucocorticoid, or other pain-relief medication
* History of daily cannabis, tobacco, or nicotine use within six months of study initiation
* BMI >30kg/m2
* Prediabetes
* Type 2 diabetes
* Health conditions that put the subject at risk to participate in exercise during this study
* Atypical or Grade 2b diabetic sensorimotor polyneuropathy
* More than one lifetime event of hospitalization for diabetic ketoacidosis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
The effect of T1D on skeletal muscle health, quantified by physiological parameters (detailed in description) | At time of study start (baseline characteristics)
  Individuals with T1D as well as their age, sex, and BMI-matched control counterparts will undergo various physiological assessments to evaluate their muscle health: strength/aerobic fitness testing, compartmental body composition assessment, blood analysis, glucose monitoring, muscle biopsy, motor neuron function evaluation, and assessments of muscle microvascular structure and function. All metrics will be compared between individuals with T1D and their non-T1D counterparts.

SECONDARY OUTCOMES:
The effect of twelve weeks of exercise on skeletal muscle health compared to baseline, quantified by physiological parameters (detailed in description) | Twelve weeks following study initiation
  Following baseline assessments, study participants will undergo a combined aerobic and resistance training program for twelve weeks. Following twelve weeks of participation in this exercise program, all study participants will undergo various physiological assessments to evaluate their muscle health: strength/aerobic fitness testing, compartmental body composition assessment, blood analysis, glucose monitoring, muscle biopsy, motor neuron function evaluation, and assessments of muscle microvascular structure and function.
The acute effect of a detraining period on skeletal muscle health compared to baseline, quantified by physiological parameters (detailed in description) | Thirteen weeks following study initiation
  Following completion of the aforementioned twelve week exercise program, study participants will undergo a seven-day detraining period consisting of unilateral knee immobilization using a hinged knee-joint immobilization brace. Immediately following this immobilization period, all study participants will undergo various physiological assessments to evaluate their muscle health: strength/aerobic fitness testing, compartmental body composition assessment, blood analysis, glucose monitoring, muscle biopsy, motor neuron function evaluation, and assessments of muscle microvascular structure and function.
The effect of a detraining period on skeletal muscle health compared to baseline, quantified by physiological parameters (detailed in description) | Seventeen weeks following study initiation
  Following completion of the aforementioned twelve week exercise program, study participants will undergo a seven-day detraining period consisting of unilateral knee immobilization using a hinged knee-joint immobilization brace. Four weeks after this immobilization period, all study participants will undergo various physiological assessments to evaluate their muscle health: strength/aerobic fitness testing, compartmental body composition assessment, blood analysis, glucose monitoring, muscle biopsy, motor neuron function evaluation, and assessments of muscle microvascular structure and function.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J Hawke, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Participant data - after deidentification.
Supporting Information: Study Protocol
Time Frame: Starting in May 2024
Access Criteria: Investigators whose proposed use of the data has been approved by an independent internal committee identified for this purpose.

REFERENCES:
- [Derived] Rebalka IA, Noguchi KS, Bulyovsky KR, Badour MI, Juracic ES, Barrett K, Brahmbhatt A, Al-Khazraji B, Punthakee Z, Perry CGR, Kumbhare DA, MacDonald MJ, Hawke TJ. Targeting skeletal muscle health with exercise in people with type 1 diabetes: A protocol for HOMET1D, a prospective observational trial with matched controls. PLoS One. 2024 May 22;19(5):e0303448. doi: 10.1371/journal.pone.0303448. eCollection 2024. PMID 38776307